CLINICAL TRIAL: NCT02960282
Title: The Role of Microbiome in Cancer Therapy
Brief Title: Gut Microbiome in Fecal Samples From Patients With Metastatic Cancer Undergoing Chemotherapy or Immunotherapy
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-16-9; NCI-2016-01584 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-16-9 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Carcinoma; Stage IV Colorectal Cancer; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer
MeSH Terms: conditions — Carcinoma; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (gut microbiome analysis): Patients undergo collection of fecal specimens at baseline, prior to start of each course of chemotherapy or immunotherapy, at the end of weeks 2, 4, 6, and 8, at the end of course 3 and courses thereafter of chemotherapy or immunotherapy, and at the time of disease progression or going off-treatment. Fecal specimens are analyzed via 16S ribosomal RNA gene sequencing, meta-transcriptomics analysis, and meta-proteomics analysis.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of fecal specimens
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies the gut microbiome in fecal samples from patients with cancer that has spread to other parts of the body who are undergoing chemotherapy or immunotherapy. Studying samples of feces from patients with metastatic cancer in the laboratory may help doctors learn if the make-up of the gut microbiome has a positive or negative influence to a patient's response to chemotherapy or immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To quantitatively determine the composition of the microflora and their gene and protein expression levels in patients with metastatic colorectal cancer being treated with fluorouracil (5-FU) based chemotherapy, or anti-PD1 immunotherapy.

SECONDARY OBJECTIVES:

I. Compare the changes in species composition and in the metabolic activities (as determined in the primary objective) with response to chemotherapy or immunotherapy.

II. Compare the changes in species composition and in the metabolic activities (as determined in the primary objective) with toxicities and side effects resulting with chemotherapy or immunotherapy.

OUTLINE:

Patients undergo collection of fecal specimens at baseline, prior to start of each course of chemotherapy or immunotherapy, at the end of weeks 2, 4, 6, and 8, at the end of course 3 and courses thereafter of chemotherapy or immunotherapy, and at the time of disease progression or going off-treatment. Fecal specimens are analyzed via 16S ribosomal ribonucleic acid (RNA) gene sequencing, meta-transcriptomics analysis, and meta-proteomics analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing and able to provide fecal samples according to protocol schedule
* COHORT A
* Diagnosis of metastatic colorectal cancer, where the metastatic disease has not been previously treated
* Scheduled to begin fluorouracil/leucovorin calcium/oxaliplatin (FOLFOX) or folinic acid-fluorouracil-irinotecan (FOLFIRI) based chemotherapy for the advanced disease
* Must have radiologic evidence of disease
* COHORT B
* Diagnosis of metastatic cancer
* Scheduled to begin pembrolizumab or another anti-PD-1 or anti-PD-L1 antibody as single agent therapy for the treatment of the advanced disease
* Must have physical or radiologic evidence of disease

Exclusion Criteria:

* Patients with a colostomy or any other issues that may prevent the standard methods for collection of stool are not eligible for this study
* Patients are not enrolled or a research protocol for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort A: Patients with metastatic colorectal cancer who will begin a FOLFOX or FOLFIRI based treatment regimen as the 1st treatment for the metastatic disease.
  Cohort B: Patients with metastatic cancer who will begin Pembrolizumab (or another anti-PD-1 or anti-PD-L1 antibody) as single agent treatment for the metastatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Best tumor response, defined as a complete response or a clear decrease in tumor burden | Up to 2 years
  The presence and amounts of species and their protocols will be compared to tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim Zandi, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States